CLINICAL TRIAL: NCT05602805
Title: Mental Health, Eating Disorders and Obesity Databank
Brief Title: BariaPSY: the Data Bank
Status: Recruiting | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Sylvain Iceta, Principal Investigator - Assistant professor, Laval University
Other Study IDs: 2023-3886, 22254
Record Dates: First submitted 2022-10-27; First posted 2022-11-02 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Bariatric Surgery Candidate; Obesity
Keywords: Obesity; Mental Health; Bariatric Surgery; Eating Disorder
MeSH Terms: conditions — Obesity; Psychological Well-Being; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Multimorbidity, the co-occurrence of several chronic conditions, is a growing phenomenon that poses new challenges for clinicians and researchers. The association between a mental health disorder and a physical health disorder represents a particularly frequent subtype of multimorbidity and is associated with greater severity and higher consumption of care. It is essential and urgent to explore the specific pathophysiology of this subtype of multimorbidity in order to develop adapted therapeutic strategies.

Psychiatric disorders, such as mood disorders, anxiety disorders, attention deficit disorder and binge eating disorder, are common in people with obesity. For example, although most of these disorders may improve after bariatric surgery, some components of these disorders, such as emotional dysregulation and impulsivity, need to be addressed as they appear to be involved in the development of addiction and suicidality after bariatric surgery. Therefore, screening and vigilance of these risks appear increasingly necessary.

To address this challenge, the BariaPsy databank aims to explore the screening of certain mental health disorders frequently observed in adults with obesity through an innovative approach that explores behaviors in the form of dimensions. It will help clinicians to quickly identify markers of certain disorders, thus helping them to further investigate the problem and provide personalized resources to their patient.

DETAILED DESCRIPTION:
The specific research objectives pursued by BariaPsy are as follows:

1. To develop a comprehensive screening tool to support the health professionals (surgeon, physician, specialized practice nurse) in their consultation regarding the mental health of the candidate for overweight or obesity management, helping them to delve deeper into the problem and to give personalized resources to their patient so that they can be well supported.
2. To evaluate the interest of such an evaluation device on the effectiveness and tolerance of the management proposed to the participants.
3. To better characterize patients with physical-mental multimorbidity and the impact of this phenotype on management, in order to issue appropriate recommendations.
4. To identify the prevalence of psychiatric disorders, including mood disorders, anxiety disorders, attention deficit disorder, and binge eating disorder, in the hospital setting, in the overweight/obese population.
5. To identify potential pathophysiological mechanisms to explain the links between mental health and obesity by relating the affected psychological dimensions to the anthropometric, metabolic and sociodemographic parameters of the participants (through information contained in the medical records).
6. Identify potential pathophysiological mechanisms to explain the links between mental health and obesity by relating the affected psychological dimensions to the parameters of current biology available in the medical record (liver, inflammatory, carbohydrate and lipid balance, etc.), but also biological and histological parameters (e.g., adipose tissue samples) in relation to the biobank or management frameworks that are already in place (e.g., in the bariatric surgery service).

Also, the participant's authorization will be requested in the Information and Consent Form to have access to their IUCPQ medical record, which contains a collection of sociodemographic, anthropometric and biological information as well as information related to their obesity management (data collection by the bariatric surgery program nurse and/or data collection carried out when the questionnaire is sent to the bariatric medicine or psychiatry programs).

The BariaPsy databank will improve the screening of certain mental health disorders frequently observed in the context of overweight or obesity in adults. The data collected will be used for several research studies with the objective of better characterizing patients with physical-mental multimorbidity and the impact of this phenotype on management, in order to issue appropriate recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Be a patient referred to the IUCPQ for management of overweight or obesity
* Have a body mass index (BMI) ≥25 kg/m2
* Be 18 years old or older

Exclusion Criteria:

* Be an incapacitated or protected adult as defined by law
* Not registered or eligible for RAMQ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred to the IUCPQ for management of overweight or obesity, thus having a body mass index (BMI) ≥25 kg/m2, and older than 18 years of age can be included in the database. This therefore implies, but is not limited to, the bariatric surgery, medicine, and psychiatry tracks of the IUCPQ. It is not necessary to have a psychiatric diagnosis according to the Diagnostic and Statistical Manual of Mental Disorders 5 (DSM-5) to be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2067-11 (Estimated); Study Completion 2072-11 (Estimated)

PRIMARY OUTCOMES:
Binge Eating Disorder (BEDS-7) | Baseline
  A screening tool that has been designed to screen adults who may have binge eating disorder.
  The results indicate whether or not the test screens for binge eating behaviors (yes or no).
Binge Eating Scale (BES) | Baseline
  To assess the presence of certain binge eating behaviors that may be indicative of an eating disorder.
  The higher the score, the more binge eating behaviors is observed. The minimum score is 0 while the maximum score is 46. The final result allows to say if the person has an absent (less than 17), moderate (between 18 and 26) or severe (more than 27) binging level.
Generalized Anxiety Disorder (GAD-7) | Baseline
  A screening tool and severity measure for generalised anxiety disorder.
  The higher the score, the higher the level of anxiety. The minimum score is 0 and the maximum score is 21. The clinically significant score is 15.
Patient Health Questionnaire (PHQ-9) | Baseline
  The PHQ-9 is a multipurpose instrument for screening, monitoring and measuring the severity of depression.
  The higher the score, the more depressive symptoms are present. The minimum score is 0 and the maximum score is 27. It allows to evaluate if there is no depression (9 and less), a major depression (between 10 and 19) or a severe major depression (20 and more).
Adult ADHD Self-Report Scale (ASRS-5) | Baseline
  To evaluate the manifestations and behaviors of attention deficit and hyperactivity disorder in adults.
  The higher the final score, the more evidence of ADHD is present. The minimum score is 6 and the maximum score is 30.
Modified Yale Food Addiction Scale 2.0 (mYFAS 2.0) | Baseline
  The mYFAS 2.0 was designed to assess food addiction using a shorter version than the YFAS 2.0.It assesses the symptoms of food addiction and the resulting distress and impaired functioning.
  The higher the level of symptoms, the more severe the food addiction. Impaired functioning and distress are scored from 0 to 2. Symptoms are scored from 0 to 11. If the functioning and distress score is 1 and above, the food addiction may be mild (2-3 symptoms), moderate (4-5 symptoms), or severe (6+ symptoms).
Impulsive Behavior Scale Short Form (UPPS-P) | Baseline
  Measurement of factors that can lead to impulsive behavior. There are five subscales: Positive Urgency, Negative Urgency, Lack of Premeditation, Lack of Perseverance, and Sensation Seeking.
  A higher score on the scale or subscale corresponds to a higher level of impulsivity. The minimum total score is 1 and the maximum total score is 4.

SECONDARY OUTCOMES:
Gender identity | Baseline (Sociodemographic Questionnaire)
  Choose from: Cisgender, Transgender, non-binary, Queer, I refuse to answer, Other
Ethnic origin | Baseline (Sociodemographic Questionnaire)
  Choose from: Black, East Asian, Latino, Middle Eastern, South Asian, Southeast Asian, South Asian descent, White, I refuse to answer, Other
Marital status | Baseline (Sociodemographic Questionnaire)
  Choose from: Single, Common-law, Married, Divorced, Widowed, I refuse to answer, Other
Highest level of education | Baseline (Sociodemographic Questionnaire)
  Choose from: None, High School, Cegep, Diploma of Vocational Studies, Vocational Technical, Undergraduate University, Graduate University, Postgraduate University or Other
Average annual income | Baseline (Sociodemographic Questionnaire)
  In dollars.
Living space for most of the year | Baseline (Sociodemographic Questionnaire)
  Choose from: House/apartment/condominium, apartment or condominium for seniors, home of a relative or friend, retirement home, adult foster home, CHSLD, other
Current employment status | Baseline (Sociodemographic Questionnaire)
  Choose from: working full time, working part time, unemployed or laid off looking for work, unemployed not looking for work, homemaker, student, retired, disable
Number of person living at your place of residence | Baseline (Sociodemographic Questionnaire)
  Choose from: living alone, 1 person, 2 persons, 3 persons, 4 persons, 5 persons or more
Weight | Baseline (Sociodemographic Questionnaire)
  In kilograms (kg).
Height | Baseline (Sociodemographic Questionnaire)
  In meters (m).
Food allergies or intolerances | Baseline (Bariatric Surgery Initial Assessment)
  Open answer
Lifestyle habits | Baseline (Bariatric Surgery Initial Assessment)
  Choice: tobacco products, electronic cigarettes (with or without nicotine), alcohol and/or drugs.
  Quantity, frequency and cessation date, if applicable, are requested.
Health history and conditions | Baseline (Bariatric Surgery Initial Assessment)
  Choice: Type 1 or 2 diabetes, hypothyroidism, hyperthyroidism, thyroid nodules, cirrhosis, inflammatory bowel disease, recent prior digestive investigation (less than 5 years), colonoscopy, abdominal surgery, bariatric surgery, other surgery, asthma, COPD, home oxygen, sleep apnea, menstruation (hysterectomy, hormone therapy, pills or IUD), coronary angioplasty (with or without stent), myocardial infarction, cardiac surgery, thrombophlebitis, coagulopathy, pulmonary embolism, renal lithiasis, CKD, psychiatric hospitalization, suicide attempt, mental health diagnosis, eating disorders, neoplasia, chronic pain, other health conditions
  If applicable, since when and followed by whom.
Family history of bariatric surgery | Baseline (Bariatric Surgery Initial Assessment)
  Open-ended questions about obesity and bariatric surgeries in the applicant's family.
Weight and diet history | Baseline (Bariatric Surgery Initial Assessment)
  Open-ended questions about current and past weight and dieting to get a sense of the person's history over time in relation to their weight.
Food history | Baseline (Bariatric Surgery Initial Assessment)
  Open-ended questions related to meal intake, meal frequency, food consumed and food-related behaviors.
Physical activity History | Baseline (Bariatric Surgery Initial Assessment)
  Open-ended questions about physical activity, which ones are practiced, how often and what barriers are encountered.
Perception of body image | Baseline (Bariatric Surgery Initial Assessment)
  Open-ended questions about body image and motivation to treat obesity.
Expectations of health care professionals | Baseline (Bariatric Surgery Initial Assessment)
  Open-ended response to know the expectations towards health professionals in the management of their obesity.
Motivation to have surgery | Baseline (Bariatric Surgery Initial Assessment)
  Since when does he want to have surgery and for what reasons?
Nutritional recommendations | Baseline (Bariatric Surgery Initial Assessment)
  Three recommendations personally issued by a nutritionist are requested.
Knowledge of bariatric surgery | Baseline (Bariatric Surgery Initial Assessment)
  Open-ended questions about the different resources that should have been consulted as well as the knowledge required (side effects, recommendations, complication and percentage of failure) are asked.

CONTACTS AND LOCATIONS:
Locations (1):
- IUCPQ, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided